CLINICAL TRIAL: NCT01202461
Title: Three-year Result of Triple Therapy of Vitrectomy, Intravitreal Triamcinolone and Macular Laser Photocoagulation for Intractable Diabetic Macular Edema
Brief Title: Triple Therapy of Pars Plana Vitrectomy and Grid/Focal Laser for Diabetic Macular Edema (DME)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Samsung Medical Center, Samsung Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-07-209
Record Dates: First submitted 2010-09-14; First posted 2010-09-15 (Estimated); Last update posted 2010-09-15 (Estimated); Status verified 2010-09

CONDITIONS: Diabetic Retinopathy; Macular Edema
Keywords: Diabetic macular edema; Combination therapy for DME; DME
MeSH Terms: conditions — Diabetic Retinopathy; Macular Edema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Triple therapy of vitrectomy, IVTA and grid/focal laser photocoagulation — all pars plana vitrectomy were accompanied with removal of retinal Internal limiting membrane (ILM) around fovea in round fashion with a dimension of approximately 2 disc diameters.
  IVTA was introduced at the end of surgery or on the next day (4mg in 0.1cc). Two weeks afterward, fluorescein angiography guided macular laser photocoagulation which consisted of direct photocoagulation on leaking microaneurysms and application of grid pattern laser was undertaken.

SUMMARY:
This study is designed to report 3-year result of triple therapy of vitrectomy, intravitreal triamcinolone and macular laser photocoagulation for intractable diabetic macular edema.

Previously author reported 1-year result(Am J Ophthalmol. 2007 Dec;144(6):878-885. Epub 2007 Oct 15.).

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of diabetes mellitus
* intractable diffuse DME (diffuse DME which did not respond to or recurred after the previous IVTA and/or macular focal laser photocoagulation)
* central subfield macular thickness (CST) greater than 250μm

Exclusion Criteria:

* presence of vitreomacular traction
* a prior history of treatment for the DME within 3 months or vitreoretinal surgery

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2010-08; Primary Completion 2010-08 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Best-corrected visual acuity | At baseline, 6,12,24,36 months after surgery
  Measurement of visual acuity at every visit. VA at every visit was compared from VA at baseline

SECONDARY OUTCOMES:
Central subfield macular thickness | 0,6,12,24,36 months after surgery
  Automatically measured central subfield thickness from Stratus OCT

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, S. Korea, South Korea